CLINICAL TRIAL: NCT02058667
Title: A Phase I Study of Twice Weekly Paclitaxel and Radical Re-irradiation Using Helical Tomotherapy for Aggressive Chest Wall Recurrences of Breast Cancer
Brief Title: Reirradiation With Concurrent Paclitaxel for Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Jonathan Michael Feddock, Principal Investigator, University of Kentucky
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-BRE-47-MCC
Record Dates: First submitted 2014-01-31; First posted 2014-02-10 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Paclitaxel; Helical Tomotherapy; Chest wall
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel+Initial Radiation+Boost (Experimental): Paclitaxel twice weekly + Initial Fields Radiation + Boost Radiation (10Gy)
  Interventions: Radiation: Paclitaxel+Initial Radiation+Boost

INTERVENTIONS:
Radiation: Paclitaxel+Initial Radiation+Boost — Paclitaxel twice weekly + Initial Fields Radiation + Boost Radiation (10Gy)

SUMMARY:
The purpose of this trial in addition to a dose finding study for concurrent Paclitaxel, will be to establish a treatment algorithm for chest wall reirradiation. A nominal margin of at least 5cm will be used on the protocol and extending it to 7cm. Considering the standard treatment of breast cancer incorporates a cumulative dose of 60Gy, delivering an additional 50.4 Gy followed by a boost should target a total dose of 120 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of breast cancer with clinical evidence of recurrent disease on the chest wall following treatment that included radiotherapy, and for which there is no current standard of care or curative resection able to be performed
* Patients are permitted to have received prior therapy, but must have received a minimum of 30 Gy to the chest wall with a minimal interval since completion of radiation therapy equal to or greater than 6 months.
* Patients are permitted to have been treated with previous systemic chemotherapy. A minimal time interval since last dose of cytotoxic chemotherapy must be equal to or greater than 21 days, and all acute toxicities should be resolved to less than grade 2, and hematologic counts should meet study criteria. With regards to toxicity, patients who have left sided chest wall recurrences should not have previously exceeded more than 450 mg/m2 doxorubicin due to expected cumulative cardiotoxicity. Prior taxane therapy is allowed, however, there should be no reported anaphylactic reactions of grade 3 or higher.
* Age ≥18 years
* ECOG performance status ≤2
* Life expectancy of greater than 3 months
* Normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin < 1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine
  * levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiotherapy within 6 months prior to entering the study or those who have not recovered to < grade 2 adverse events due to radiation
* Patients who have experienced a previous grade 3 or 4 anaphylactic reaction to Paclitaxel.
* Patients with grade > 2 neuropathy attributable to previous administration of Taxane chemotherapy.
* Patients who have received prior chemotherapy are allowed, provided they have been off systemic therapy for 21 days and all acute toxicities have resolved to less than grade 2. Patients who have received Paclitaxel within 3 months of study entry and have developed documented progressive disease despite therapy.
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should have their brain metastases treated prior to enrollment on this protocol. Subjects may enroll on this trial after completion of whole brain radiation therapy and/or Stereotactic Radiosurgery, provided they are clinically without evidence of progressive brain metastases.
* Patient who are actively receiving other cytotoxic or antibiologic chemotherapies. For patients with Her-2/neu positive disease, Trastuzumab (Herceptin) is NOT ALLOWED on this study, and should be withheld during the 8 weeks of therapy, and can be resumed no sooner than 14 days following completion of protocol therapy
* Women with a confirmed intrauterine pregnancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Paclitaxel is an antimicrotubule agent with known potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Paclitaxel, breastfeeding should be discontinued if the mother is treated with Paclitaxel
* HIV-positive patients on combination antiretroviral therapy are ineligible.
* Patients with poor cardiac function defined as an ejection fraction (EF) < 40% are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
MTD identification | From first dose at week 1 until unacceptable toxicity occurs, up to 7 weeks
  To identify the maximum tolerated dose of twice weekly Paclitaxel given concurrently with chest wall re-irradiation using helical tomotherapy for aggressive breast cancer recurrences

SECONDARY OUTCOMES:
Time to progression | Up to 6 months
Local Control Rate of Dermal Disease at 6 months | 6 months
Rate of study-defined grade 1-2 toxicities, and all grade 3 or higher toxicities | Up to 6 months
Her-2/neu transformation | 1-6 months
  Her-2/neu transformation from initial therapy to the time of development of dermal metastasis or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Feddock, MD, Principal Investigator — UK Markey Cancer Center
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States